CLINICAL TRIAL: NCT02401763
Title: Investigating the Role of Mucin and Mucin Glycosylating Enzymes in Nasopharyngeal Carcinoma and Salivary Gland Cancer and Their Correlation With Clinical Prognosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412126RIND
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Salivary Gland Cancer; Nasopharyngeal Carcinoma
Keywords: biomarker
MeSH Terms: conditions — Salivary Gland Neoplasms; Nasopharyngeal Carcinoma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nasopharyngeal carcinoma and salivary gland tumor: patients diagnosed and treated in National Taiwan University Hospital

SUMMARY:
Nasopharyngeal carcinoma (NPC) is the tenth leading cancers in Taiwan and investigating its biomarker is important for understanding the mechanism of its pathogenesis.

DETAILED DESCRIPTION:
NPC is the tenth leading cancers in Taiwan and investigating its biomarker is important for understanding the mechanism of its pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* NPC and salivary gland tumor diagnosed and treated in HTUH

Exclusion Criteria:

* previous treatment or surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPC and salivary gland tumor diagnosed and treated in HTUH
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The difference of expression level of mucin glycosylating enzymes (by immunohistochemistry) in nasopharyngeal carcinoma and salivary gland tissues | 1~5 years after patients received definite therapy

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, Principal Investigator — NTUH